CLINICAL TRIAL: NCT05454085
Title: Could Bisphenol-A Have a Role in the Etiology of Neural Tube Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Collaborators: Bursa Yuksek Ihtisas Education and Research Hospital (Unknown)
Responsible Party: Principal Investigator, Nefise Nazlı YENIGUL, Ph.D. Associet Professor Department of Obstetrics and Gynecology, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021/02-12
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Neural Tube Defects; Bisphenol-A
Keywords: Bisfenol A; amniocentesis; neural tube defect
MeSH Terms: conditions — Neural Tube Defects | interventions — Bisphenols

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pregnancies with neural tube defects (Other): patients with pre-diagnosis of neural tube defects (47 patients).
  Interventions: Dietary Supplement: Bisphenol-A
- pregnancies without neural tube defects (Other): patients with abnormal maternal serum screening test or prenatal diagnosis test, patients with abnormal ultrasonography findings (45 patients)
  Interventions: Dietary Supplement: Bisphenol-A

INTERVENTIONS:
Dietary Supplement: Bisphenol-A — measurement of BPA levels in maternal blood and amniotic fluid

SUMMARY:
Our aim in this study is in patients with a diagnosis of neural tube defect; is the measurement of BPA levels in maternal blood and amniotic fluid.

DETAILED DESCRIPTION:
This prospective observational study was conducted with 92 patients aged 18 - 45 years who had amniocentesis at 15 - 22 weeks of gestation at Bursa Yüksek İhtisas Training and Research Hospital between April 15, 2021 and April 15, 2022. Patients were divided into two groups according to amniocentesis indications. Group 1: patients with abnormal maternal serum screening test or prenatal diagnosis test, patients with abnormal ultrasonography findings (45 patients), Group 2: patients with pre-diagnosis of NTD (47 patients). During the amniocentesis procedure, the first 5cc amniotic fluid and maternal serum samples were collected from the patients. The obtained samples were stored at -80°C until the end of the study. After all samples were collected, BPA values were measured by ELISA method.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a single pregnancy, had a pre-diagnosis of neural tube defect or had amniocentesis between 15 and 22 weeks of age with other indications
* patients had an uncomplicated pregnancy before the procedure
* patients had no vaginal infection

Exclusion Criteria:

* Multiple pregnancies,
* pregnant women who developed complications due to amniocentesis
* pregnant women with known infective or autoimmune diseases before pregnancy
* those whose spouses or themselves worked in the plastics industry
* patients who could not obtain enough amniotic fluid despite meeting the study criteria during the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
BPA levels | 1 year
  measurement of BPA levels in maternal blood and amniotic fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı YENIGUL, Bursa, Turkey (Türkiye)